CLINICAL TRIAL: NCT04177368
Title: Nutritional Assessment of Children With End Stage Renel Disease(ESRD) on Regular Hemodialysis
Brief Title: Nutritional Assessment of Children With ESRD on Dialysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, shimaa kamel ahmed, principle investigator, Assiut University
Other Study IDs: NACWESRD
Record Dates: First submitted 2018-09-22; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Assessment of Nutrition in ESRD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- assess nutrition with regular dialysis: This study aims to assess the growth and the nutritional status in children with end-stage kidney disease on regular hemodialysis to define the degree of malnutrition , predict and quantify the risk for complications deriving from impaired nutritional status .Giving them theragran 60ml ,twice daily for 3 month.
  Interventions: Dietary Supplement: Theragran 60ml

INTERVENTIONS:
Dietary Supplement: Theragran 60ml — history,examination and biochemical values

SUMMARY:
Normal growth can be divided into four important phases: prenatal, infantile, childhood and pubertal. Nutrition is important at all phases of growth, but particularly so during the infantile phase because the rate of growth is higher than at any other time of life and is less dependent on growth hormone than during other phases. During the childhood phase, growth becomes more dependent on the GH/insulin-like growth factor-1 axis; growth rate decelerates continuously until the pubertal phase. The pubertal phase results from the coordination of GH and sex steroid production. Together they have an anabolic effect on muscle mass, bone mineralization and body proportions. It is another phase of rapid growth so that nutrition can again modify the genetic growth potential.

DETAILED DESCRIPTION:
Achieving an optimal nutritional status is essential for managing paediatric chronic kidney disease, and dietary guidance is frequently provided in clinical practice to achieve a metabolic balance, which is vital for normal growth. Guidelines addressing optimal macro- and micronutrient intake for children with CKD are available, with intake of sodium, potassium, phosphorus, protein, and total calories being common targets of nutritional monitoring.

Normal nutrition can be defined as maintenance of normal growth and body composition. Although it is agreed that nutritional assessment is important in chronic renal failure, there is no single or easy definition or measure of inadequate nutritional status: measurement of nutritional parameters are complicated in CRF because of salt and water imbalances and the potential inappropriateness of using age matched controls in a population that is short and may be delayed in puberty; it has been suggested that it is more appropriate, therefore, to express measures relative to height age and/or pubertal stage.

Malnutrition is common in hem dialysis patients and is a powerful predictor of morbidity and mortality. Although much progress has been made in recent years in identifying the causes and pathogenesis of malnutrition in hemodialysis patients, as well as recognizing the link between malnutrition and morbidity and mortality, no consensus has been reached concerning its management. Along with such conventional interventions as nutritional counseling, oral nutritional supplements, and dialectic parental nutrition, novel preventive and therapeutic strategies have been tested, such as appetite stimulants, growth hormone, androgenic anabolic steroids, and anti-inflammatory drugs, with contradictory and non conclusive results. Malnutrition still remains a great challenge for nephrologists in the third millennium.

Growth failure is almost inextricably linked with chronic kidney disease and end-stage renal disease.Growth failure in CKD has been associated with both morbidly and mortality .Growth failure in the setting of kidney disease is multi factorial and is related to poor nutritional status as well as co morbidities ,such as anemia, bone and mineral disorders, and alterations in hormonal responses, as well as to aspects of treatment such as steroid exposure. Initial reports of renal dwarfism date back to the turn of the twentieth century. Despite advances in conservative treatment and renal replacement therapies, 30-60% of patients with ESRD are short at adulthood.

Hypoalbuminemia is the most powerful predictor of mortality in end-stage renal disease. Since protein-calorie malnutrition can decrease albumin synthesis it is assumed that hypoalbu minemia results principally from malnutrition in these patients, but albumin synthesis may also be decreased as part of the acute-phase response, and hypoalbuminemia can also result from redistribution of albumin pools or from albumin losses.Serum albumin has been identified as a surrogate marker for nutritional status and morbidity / mortality in patients with end-stage renal failure. Although serum albumin may be a reflection of nutrition, low levels may be due to haemodilution, nephrotic syndrome or chronic infection / inflammation.

The most commonly used assessment of nutrition is height and weight, along with head circumference in younger children, plotted on percentile charts. Another way of expressing the relative weight and height is the body mass index, which is important because extremes are associated with increased morbidity and mortality. Skin fold thickness is a measure of subcutaneous fat and mid-arm circumference is a reflection of muscle mass and may therefore be more useful in determining body composition than the calculation of BMI alone.

ELIGIBILITY:
Inclusion Criteria:

* Age : 5-15 Years
* Sex : Male & Female
* Diagnosed as ESRD and on regular hemodialysis.
* Estimated glomerular filtration rate (eGFR): greater than or equal to 5 mL/min and less than or equal to 15 mL/min.
* Clinically stable.

Exclusion Criteria:

* • Infants & adults

  * Not expected to initiate dialysis
  * Estimated glomerular filtration rate (eGFR): greater than or equal to 15 mL/min and less than or equal to 60 mL/min.
  * Clinically unstable

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: assess nutrition with regular dialysis This study aims to assess the growth and the nutritional status in children with end-stage kidney disease on regular hemodialysis to define the degree of malnutrition , predict and quantify the risk for complications deriving from impaired nutritional status .Giving them theragran 60ml ,twice daily for 3 month.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
prevention of malnutrition in children on regular dialysis | 1 year
  malnutrion can be preventable by good nutrition assessment

CONTACTS AND LOCATIONS:
Overall Officials: Shimaa Kamel Ahmed, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided
No Plan till this time